CLINICAL TRIAL: NCT04318561
Title: A Prospective, Randomized, Double-blinded Study to Evaluate the Safety, Biodistribution, Dosimetry and Lesion Detection Ability of Gallium-68 Labeled LM3 for the Diagnostic Imaging of Metastatic, Well-differentiated Neuroendocrine Tumors Using PET/CT
Brief Title: Gallium-68 Labeled LM3 PET/CT in Neuroendocrine Tumors
Acronym: PET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LM3NT
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The details of patient groups will be sealed in sequentially numbered, opaque, sealed envelopes generated by Xuezhu Wang from the nuclear medicine department, Peking Union Medical College Hospital, who will not participate in other parts of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gallium-68 NODAGA-LM3 group (Experimental): Patients will undergo a Gallium-68 NODAGA-LM3 PET/CT as well as a Gallium-68 DOTATATE PET/CT.
  Interventions: Diagnostic Test: Gallium-68 NODAGA-LM3 PET/CT; Diagnostic Test: Gallium-68 DOTATATE PET/CT
- Gallium-68 DOTA-LM3 group (Experimental): Patients will undergo a Gallium-68 DOTA-LM3 PET/CT as well as a Gallium-68 DOTATATE PET/CT.
  Interventions: Diagnostic Test: Gallium-68 DOTA-LM3 PET/CT; Diagnostic Test: Gallium-68 DOTATATE PET/CT

INTERVENTIONS:
Diagnostic Test: Gallium-68 NODAGA-LM3 PET/CT — Twenty patients will take this intervention. They will be further divided into two sub-groups with the same interventional radiopharmaceutical (Gallium-68 NODAGA-LM3) but different scanning protocols (Protocol A and Protocol B). The first enrolled 8 patients will go with Protocol A, who will undergo serial whole-body PET/CT scans at multiple time points (5m, 10m, 20m, 40m, 1h, 2h) after administering 40ug/150-200MBq Gallium-68 NODAGA-LM3. Baseline safety assessment will be conducted right before the study. The following 12 patients will go with Protocol B, who will undergo a whole-body PET/CT scan at 1 hour after administering 40ug/150-200MBq Gallium-68 NODAGA-LM3.
  Arms: Gallium-68 NODAGA-LM3 group
Diagnostic Test: Gallium-68 DOTA-LM3 PET/CT — Twenty patients will take this intervention. They will be further divided into two sub-groups with the same intervention radiopharmaceutical (Gallium-68 DOTA-LM3) but different scanning protocols (Protocol C and Protocol D). The first enrolled 8 patients will go with Protocol C, who will undergo serial whole-body PET/CT scans at multiple time points (5m, 10m, 20m, 40m, 1h, 2h) after administering 40ug/150-200MBq Gallium-68 DOTA-LM3. Baseline safety assessment will be conducted right before the study. The following 12 patients will go with Protocol D, who will undergo a whole-body PET/CT scan at 1 hour after administering 40ug/150-200MBq Gallium-68 DOTA-LM3.
  Arms: Gallium-68 DOTA-LM3 group
Diagnostic Test: Gallium-68 DOTATATE PET/CT — All patients have to do a Gallium-68 DOTATATE PET/CT scan (40ug/150-200MBq, 1h post-injection) for comparison on the next day of LM3 scan. Safety assessment and tolerability of the previous LM3 study will be conducted right before the study.

SUMMARY:
LM3 is a novel somatostatin receptor antagonist, while Gallium-68 DOTATATE is a typical somatostatin receptor agonist, This study is to evaluate the safety, biodistribution, dosimetry, and lesion detection ability of Gallium-68 labeled somatostatin receptor antagonist LM3 for the diagnostic imaging of metastatic, well-differentiated neuroendocrine tumors using positron emission tomography / computed tomography (PET/CT).

The results will be compared between antagonist Gallium-68 labeled LM3 and agonist Gallium-labeled DOTATATE in the same group of patients.

It will also be compared between the two different antagonists, Gallium-68 DOTA-LM3 and Gallium-68 NODAGA-LM3, in two parallel-designed arms.

DETAILED DESCRIPTION:
Patients with histologically confirmed metastatic, well-differentiated neuroendocrine tumors will be recruited in this study.

All patients will be randomized into two groups: Gallium-68 NODAGA-LM3 group and Gallium-68 DOTA-LM3 group.

The study will be divided into the following 2 parts:

Part ONE, which will enroll 16 patients (8 in each group), focuses on the safety evaluation, biodistribution, and dosimetry. In Part A, patients will undergo serial whole-body PET/CT scans at multiple time points (5m, 10m, 20m, 40m, 1h, 2h) after administering 40ug/150-200MBq Gallium-68 NODAGA-LM3 or Gallium-68 DOTA-LM3 (according to their group).

Part TWO, which will enroll 24 patients (12 in each group) and follows Part A study, focuses on lesion detection ability. In Part B, patients will undergo one whole-body PET/CT scan at 1 hour after administering 40ug/150-200MBq Gallium-68 NODAGA-LM3 or Gallium-68 DOTA-LM3 (according to their group).

All patients need to do a Gallium-68 DOTATATE PET/CT scan (40ug/150-200MBq, 1h post-injection) for comparison on the next day.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients of either gender, aged ≥ 18 years.
* Histologically confirmed diagnosis of Metastatic, well-differentiated neuroendocrine tumor.
* A diagnostic computed tomography (CT) or magnetic resonance imaging (MRI) of the tumor region within the previous 6 months prior to dosing day is available.
* At least 1 measurable lesion based on RECIST v1.1.
* Blood test results as follows (White blood cell: ≥ 3*10^9/L, Hemoglobin: ≥ 8.0 g/dL, Platelets: ≥ 50x10^9/L, Alanine aminotransferase / Aspartate aminotransferase / Alkaline phosphatase: ≤ 5 times upper limit od normal (ULN), Bilirubin: ≤ 3 times ULN)
* Serum creatinine: within normal limits or < 120 μmol/L for patients aged 60 years or older.
* Calculated Glomerular filtration rate (GFR) ≥ 45 mL/min.

Exclusion Criteria:

* Known hypersensitivity to Gallium-68, to NODAGA, to DOTA, to LM3, to TATE or to any of the excipients of Gallium-68 DOTA-LM3, Gallium-68 NODAGA-LM3 or Gallium-68 DOTATATE.
* Presence of active infection at screening or history of serious infection within the previous 6 weeks.
* Therapeutic use of any somatostatin analog, including long-acting Sandostatin (within 28 days) and short-acting Sandostatin (within 2 days) prior to study imaging. If a patient is on long-acting Sandostatina, then a wash-out phase of 28 days is required before the injection of the study drug. If a patient is on short-acting Sandostatin, then a wash-out phase of 2 days is required before the injection of the study drug.
* Any neuroendocrine tumor-specific treatment between antagonist and agonist scans.
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study.
* Pregnant or breast-feeding women.
* Current history of any malignancy other than neuroendocrine tumor; patients with a secondary tumor in remission of > 5 years can be included.
* Any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure[Safety and tolerability] | Within 1 hour prior to the administration of radiopharmaceuticals.
  Measured in millimetre of mercury.
Heart rate[Safety and tolerability] | Within 1 hour prior to the administration of radiopharmaceuticals.
  Measured in beats per minute.
Pulse oximetry[Safety and tolerability] | Within 1 hour prior to the administration of radiopharmaceuticals.
  Measured in percentage.
Electrocardiogram QT interval[Safety and tolerability] | Within 1 hour prior to the administration of radiopharmaceuticals.
  3-lead electrocardiogram
Incidence of adverse effect[Safety and tolerability] | From right after tracer injection to 24-hours post-injection
  According to version 4.03 of the Common Terminology Criteria for Adverse Events.

SECONDARY OUTCOMES:
Cmax (maximum concentration achieved in units of Bq/ml) | From right after tracer injection to 2-hours post-injection
  Determination of Cmax for target lesion and discernible organs
Tmax (time to achieve Cmax) | From right after tracer injection to 2-hours post-injection
  Determination of Tmax for target lesion and discernible organs.
Standard uptake value (SUV) | From right after tracer injection to 2-hours post-injection
  Determination of SUV for detected lesions and discernible organs of 68Ga-DOTA-LM3, 68Ga-NODAGA-LM3, and 68Ga-DOTATATE scan.
Lesion numbers | From right after tracer injection to 2-hours post-injection
  Determination of lesion numbers of 68Ga-DOTA-LM3, 68Ga-NODAGA-LM3, and 68Ga-DOTATATE scan.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjia Zhu, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu W, Jia R, Yang Q, Cheng Y, Zhao H, Bai C, Xu J, Yao S, Huo L. A prospective randomized, double-blind study to evaluate the diagnostic efficacy of 68Ga-NODAGA-LM3 and 68Ga-DOTA-LM3 in patients with well-differentiated neuroendocrine tumors: compared with 68Ga-DOTATATE. Eur J Nucl Med Mol Imaging. 2022 Apr;49(5):1613-1622. doi: 10.1007/s00259-021-05512-y. Epub 2021 Dec 7. PMID 34874478